CLINICAL TRIAL: NCT07069634
Title: The Effect of Individualised Education Using the Teach Back Method on Depression Levels in Hemodialysis Patients
Brief Title: Teach Back Method on Depression Levels in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Büşra Zehra BÜYÜKKILIÇ, Research Assistant, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BUYUKKILIC
Record Dates: First submitted 2025-06-23; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Hemodialysis Patients; Teach Back; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: The research is a two-center, randomized, interventional (educational) type research with intervention and control groups, pre-test-post-test design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): They were asked to respond to the scale questions (post-test) 12 weeks after the pre-test and the first interview at the beginning of the study.
- Individual training using the Teach Back Method (Experimental): Pre-test was collected with patients receiving hemodialysis treatment. Individual training was given to the intervention group patients using the Tell What You Learned Method using face-to-face and individual interview techniques. The training was carried out in 3 sessions. After the training sessions were completed, they were asked to answer questions asked by the researcher in order to evaluate their knowledge, skills and behaviors regarding the Tell What You Learned Method. The intervention group patients were given a post-test in the third month (12th week) after the first interview.
  Interventions: Other: Individual training using the Teach Back Method

INTERVENTIONS:
Other: Individual training using the Teach Back Method — Day 1 (Monday): Patients are introduced to the study; consent forms are signed, and initial forms are completed. An educational booklet is provided and explained. General information about hemodialysis and treatment is delivered using the Teach-Back Method.
  Day 2 (Wednesday): Patients recall previous session topics; unclear points are clarified. Education focuses on fluid and dietary restrictions and the importance of adherence, using the Teach-Back Method.
  Day 3 (Friday): Patients summarize previous content; the researcher reinforces unclear areas. Education covers medication adherence and lifestyle habits, again using the Teach-Back Method.
  Arms: Individual training using the Teach Back Method

SUMMARY:
Background: Depression is one of the most common psychiatric disorders among hemodialysis patients and is associated with increased morbidity and mortality. Due to the chronic nature of the disease and the burdens of treatment, patients often experience psychological distress. The Teach-Back Method is a patient education strategy that ensures comprehension and retention by having patients repeat the information in their own words, and has shown promise in managing chronic conditions.

Objective: This study aimed to evaluate the effect of individualized education using the Teach-Back Method on the depression levels of adult patients undergoing hemodialysis.

Methods: This was a two-center, randomized controlled interventional study with a pre-test-post-test design. A total of 40 patients with End-Stage Renal Disease (ESRD), aged between 18-65, who had been receiving hemodialysis for at least three months, were randomly assigned to intervention (n=20) and control (n=20) groups. The intervention group received three sessions of individualized education using the Teach-Back Method, while the control group received no intervention during the study. Depression levels were assessed using the Beck Depression Inventory (BDI) before and three months after the intervention.

Hypothesis

H1: Individual education provided using the Teach-Back Method reduces the level of depression in adult ESRD patients receiving hemodialysis treatment.

ELIGIBILITY:
Inclusion Criteria:

* Those who have been diagnosed with end-stage renal failure and have received hemodialysis treatment 3 times a week for 4 hours for at least 3 months, have no communication problems and are between the ages of 18-65

Exclusion Criteria:

* Patients who did not attend any of the educational sessions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Depression scores | For 12 weeks The intervention group consisted of patients who received hemodialysis treatment on Tuesdays, Thursdays, and Saturdays, and the control group consisted of patients who received treatment on Mondays, Wednesdays, and Fridays.
  Individual education given to adult ESRD patients receiving hemodialysis using the TeachBack Method reduces depression levels.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Faculty of Nursing, Istanbul, Istanbul, Turkey (Türkiye)